CLINICAL TRIAL: NCT04259411
Title: A Prospective, Multi-Center, Single-Arm, Post Market Study of the MitraClip System for the Treatment of Symptomatic Mitral Regurgitation in China
Brief Title: MitraClip China PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10263
Record Dates: First submitted 2019-09-23; First posted 2020-02-06 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Mitral Regurgitation
Keywords: MR; Mitral Regurgitation; MitraClip
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- MitraClip (Experimental): Subject will receive MitraClip procedure with MitraClip NTR System or MitraClip XTR System.
  Interventions: Device: MitraClip procedure

INTERVENTIONS:
Device: MitraClip procedure — MitraClip procedure with MitraClip NTR System or MitraClip XTR System

SUMMARY:
The MitraClip System is the first commercially available catheter-based option for the treatment of MR. The MitraClip System was developed as an alternate percutaneous technology which may serve as a viable therapeutic option for open-heart surgery. Treatment with the MitraClip device allows patients to undergo a less invasive procedure that can mechanistically reduce MR and allow for improved quality of life. The MitraClip procedure is performed under general anesthesia without the use of a heart-lung machine, with recovery typically lasting two to three days.

DETAILED DESCRIPTION:
Mitral regurgitation (MR) is the most common heart valve condition in the world. MR occurs when the mitral valve does not close properly, allowing blood to leak back into the upper chamber of the heart. As a result, the heart may try to pump harder in order to compensate for the decrease in blood flow to the rest of the body. Patients with severe MR suffer from debilitating symptoms such as shortness of breath, heart palpitations, lightheadedness, and fatigue. These patients are at risk of poor quality of life, marked limitation in activity, repeated heart failure hospitalizations, and increased mortality. Chronic severe MR is often associated with heart failure and can lead to death if left untreated.

While mitral valve repair or replacement surgery is currently regarded as standard of care, many patients with clinically significant MR are at an unacceptable risk of morbidity and mortality and are therefore not appropriate surgical candidates. To optimize afterload reduction and treatment of fluid load, these patients are often treated with medical management (i.e., beta blockers, ACE inhibitors, angiotensin II receptor blockers) which may relieve MR symptoms, but does not address the underlying cause of the condition. As a result, a significant portion of patients treated medically continue to progress to heart failure and experience an increasingly debilitating quality of life. A significant unmet clinical need thus exists for the treatment of moderate-to-severe and severe MR in high surgical risk patients.

The MitraClip System has been in clinical use for treatment of significant MR since 2003. The MitraClip System received CE (Conformité Européenne) Mark for both DMR and FMR indications in March 2008 and was approved by FDA for DMR indication in October 2013 and for FMR indication in March 2019. The system is approved for use in more than 102 countries or regions worldwide. More than 100,000 patients have undergone the MitraClip procedure worldwide. On June 15, 2020, the MitraClip System has been approved for clinical use in China.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects is eligible to receive the MitraClip per the current approved MitraClip System IFU. (If any update or amendment on the IFU, the latest version of IFU shall be followed.)
2. Subject is 18 years-old or above.
3. Subjects who give consent for study procedure.

Exclusion Criteria:

1. Subject cannot tolerate procedural anticoagulation or anti-platelet regimen.
2. Subject with active endocarditis of mitral valve.
3. Subject with rheumatic mitral valve disease.
4. Subject with echocardiographic evidence of intracardiac, IVC or femoral venous thrombus.
5. Subject is unlikely to survive the protocol follow up period of 12-months after device implant.
6. Subject has insufficient or lost ability to maintain their will and rights.
7. Subject is illiterate.
8. Pregnant or nursing subjects and those who plan pregnancy during the study follow-up period
9. Subject participates in another clinical study that may impact the follow-up or results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2025-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle J Brunner, Study Director — Abbott Structural Heart
Locations (5):
- China (5):
  - Fuwai Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen, Fujian
  - Fuwai Hospital Chinese Academy of Medical Sciences, Shenzhen, Shenzhen, Guangdong
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The 2nd Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total 51 subjects were enrolled across five investigational sites between December 6, 2021, and April 15th, 2024 and follow-up at discharge, 30 days and 1 year.
Period: Overall Study
Arm/Group | MitraClip
Started | 51
30 days | 49
1 year | 48
Completed | 48
Not Completed | 3
Not completed — Death | 1
Not completed — Missed visit | 2

BASELINE CHARACTERISTICS:
Arm/Group | MitraClip
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 51
Weight [Mean (Standard Deviation); unit: kg] | 60.2 (13.8)
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 22.6 (4.1)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 74.1 (12.7)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 120.2 (19.7)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 69.9 (11.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Acute Procedural Success (APS)
Description: APS is defined as successful implantation of the MitraClip device(s) with resulting MR severity of 2+ or less as determined by the ECL assessment of a discharge echocardiogram (30-day echocardiogram will be used if discharge echocardiogram is unavailable or uninterpretable).
Time Frame: Discharge/30days
Population: The analysis population included all eligible and consented subjects implanted with a MitraClip device. The TTE images at discharge and 30 days were not evaluable by the echo core lab in 2 subjects, hence APS was evaluable for 49 subjects
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip
Number analyzed (Participants) | 49
percentage of participants | 93.9

2. Primary Outcome: Percentage of Participants With Freedom From Major Adverse Event (MAE)
Description: A Major Adverse Event (MAE) was determined as the composite of death, stroke, myocardial infarction (MI), renal failure, and non-elective cardiovascular surgery for device- or procedure-related adverse events occurring after the femoral vein puncture for transseptal access.
Time Frame: 30 days
Population: The analysis population included all eligible and consented subjects implanted with a MitraClip device.
Measure: Number; unit: percentage of participants
Arm/Group | MitraClip
Number analyzed (Participants) | 51
percentage of participants | 100.0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | MitraClip
All-Cause Mortality (participants affected / at risk) | 1/51
Serious Adverse Events (participants affected / at risk) | 16/51
Other Adverse Events (participants affected / at risk) | 25/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MitraClip (N=51)
Arrhythmia (Cardiac disorders) | 2
Atrial Fibrillation (Cardiac disorders) | 3
Cardiac Arrest (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 3
Cardiac Failure Chronic (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 2
Left Ventricular Failure (Cardiac disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1
Inguinal Hernia (Gastrointestinal disorders) | 1
Large Intestine Polyp (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Covid-19 (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1
Electrolyte Imbalance (Metabolism and nutrition disorders) | 2
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 2
Chronic Kidney Disease (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Aortic Aneurysm Repair (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MitraClip (N=51)
Anemia (Blood and lymphatic system disorders) | 6
Mitral Valve Incompetence (Cardiac disorders) | 4
Tricuspid Valve Incompetence (Cardiac disorders) | 1
Thyroid Mass (Endocrine disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 1
Chronic Gastritis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Functional Gastrointestinal Disorder (Gastrointestinal disorders) | 1
Chest Pain (General disorders) | 2
Decreased Activity (General disorders) | 1
Hypothermia (General disorders) | 1
Hepatic Failure (General disorders) | 1
Bronchitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Post Procedural Infection (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 3
Upper Respiratory Tract Infection (Infections and infestations) | 3
Urinary Tract Infection Enterococcal (Infections and infestations) | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1
Subdural Hematoma (Injury, poisoning and procedural complications) | 1
Weight Decreased (Investigations) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 2
Hypoproteinemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Carotid Arteriosclerosis (Nervous system disorders) | 1
Lacunar Infarction (Nervous system disorders) | 1
Transient Ischemic Attack (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Hydronephrosis (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 2
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Calcification (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 2
Hemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the earliest of: Sponsor's Study Results Disclosure; or 12 months after study completion or termination at all sites, PI shall publish results. PI shall provide Sponsor, 60 days before submission for publication, with a draft to ascertain if patentable subject matter or Sponsor Confidential Information are disclosed. Sponsor shall return comments to PI within 60 days after receipt of draft. PI shall delay publication another 60 days if Sponsor requests for proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT04259411/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT04259411/SAP_001.pdf